CLINICAL TRIAL: NCT07020065
Title: Reduced-dose Carboplatin-doublet-chemotherapy + Cemiplimab vs Cemiplimab Monotherapy in Treatment Naive Older and Frail Patients With Metastatic NSCLC With PD-L1 <50% A Multicentre Randomized Open-label Phase II Trial
Brief Title: Reduced-dose Carboplatin-doublet-chemotherapy + Cemiplimab vs Cemiplimab Monotherapy in Treatment Naive Older and Frail Patients With Metastatic NSCLC With PD-L1 <50%
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 18/24
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic NSCLC - Non-Small Cell Lung Cancer
Keywords: Reduced-dose chemotherapy; Cemiplimab; carboplatin; metastatic NSCLC; PD-L1 <50%; Non-Small Cell Lung Cancer; older and frail patients; phase II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab; Carboplatin; Pemetrexed; Gemcitabine; Paclitaxel

STUDY DESIGN:
Intervention Model Description: A multicenter randomized open-label phase II trial, with parallel design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Non-squamous histology:
  * carboplatin IV AUC 3 day 1
  * pemetrexed IV 300 mg/m2 day 1
  * cemiplimab IV 350 mg, day 1 Every 3 weeks, for 4 cycles, followed by maintenance treatment with cemiplimab with or without pemetrexed (at same dose and interval as above).
  Squamous histology:
  * carboplatin IV AUC 1.5 day 1, d8
  * gemcitabine IV 600 mg/m2 day 1, d8
  * cemiplimab IV 350 mg, day 1 Every 3 weeks, for 4 cycles, followed by maintenance treatment with cemiplimab (350 mg q3w)
  Any histology:
  * carboplatin IV AUC 1.5 day 1, d8
  * paclitaxel IV 50 mg/m2 day 1, d8
  * cemiplimab IV 350 mg, day 1 Every 3 weeks, for 4 cycles, followed by maintenance treatment with cemiplimab (350 mg q3w)
  Interventions: Drug: Cemiplimab; Drug: Carboplatin; Drug: Pemetrexed & Gemcitabine; Drug: Paclitaxel
- Comparator arm (Active Comparator): cemiplimab IV 350 mg, day 1 Every 3 weeks (max. 2 years)
  Interventions: Drug: Cemiplimab

INTERVENTIONS:
Drug: Cemiplimab — cemiplimab IV 350 mg, day 1
Drug: Carboplatin — carboplatin IV AUC 3 day 1
  Arms: Experimental arm
Drug: Pemetrexed & Gemcitabine — pemetrexed IV 300 mg/m2 day 1 gemcitabine IV 600 mg/m2 day 1, d8
  Arms: Experimental arm
Drug: Paclitaxel — paclitaxel IV 50 mg/m2 day 1, d8
  Arms: Experimental arm

SUMMARY:
Metastatic non-small cell lung cancer is often treated with a combination of chemotherapy and immunotherapy. In patients over the age of 70, some are already in poor health and frail, requiring assistance with daily activities, for example. Older and/or frail individuals often do not tolerate standard-dose chemotherapy well, and their risk of side effects is higher than that of younger patients.

For this reason, the SAKK 18/24 study is investigating how effective and safe chemotherapy is in patients over 70 years of age when the chemotherapy drugs are administered at lower doses than usual. The aim of the study is to find a potentially effective and well-tolerated treatment for older people with metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
This randomized, open-label, phase II clinical trial evaluates the efficacy, safety, and overall treatment utility of reduced-dose platinum-doublet chemotherapy (rdCT) in combination with cemiplimab (cemi) versus cemiplimab monotherapy in older and/or frail patients with stage III/IV non-small cell lung cancer (NSCLC) and PD-L1 expression <50%. The study specifically addresses a major evidence gap for a vulnerable patient population often underrepresented in registrational trials.

Cemiplimab in combination with full-dose carboplatin-based doublet chemotherapy is a Swissmedic-approved first-line treatment for advanced NSCLC, based on data from EMPOWER-Lung 03. However, full-dose chemotherapy regimens (e.g., carboplatin AUC 5 + pemetrexed, paclitaxel, or gemcitabine) are frequently associated with prohibitive toxicity in elderly and/or frail patients. Over half of all newly diagnosed mNSCLC cases occur in individuals aged 70 or older, many of whom present with frailty or multimorbidity. While atezolizumab monotherapy has shown a survival benefit over single-agent chemotherapy in older, treatment-ineligible patients (IPSOS trial), overall outcomes remain suboptimal.

In clinical practice, rdCT regimens are commonly used in this patient population, despite limited prospective evidence. The present study uses the G8 screening tool-a validated geriatric assessment instrument-to identify patients at risk for increased treatment toxicity and to support treatment adaptation.

Objectives The primary objective is to compare overall survival (OS) between rdCT + cemiplimab and cemiplimab monotherapy. Secondary objectives include comparison of progression-free survival (PFS), objective response rate (ORR), adverse events (AE), health-related quality of life (HRQoL), and overall treatment utility (OTU).

Design and Interventions This is a multicenter, randomized, open-label, parallel-group study enrolling approximately 156 patients (78 per arm) across ~17 sites in Switzerland. Eligible patients are ≥70 years old, have a G8 score ≤14 or are deemed unsuitable for full-dose chemotherapy, and have advanced or metastatic NSCLC without actionable genomic alterations and PD-L1 <50%.

Patients are randomized to one of two arms:

* Experimental Arm: rdCT + cemiplimab
* Control Arm: cemiplimab monotherapy Patients who progress and are deemed suitable may cross over to receive rdCT + cemiplimab.

Cemiplimab maintenance continues until disease progression, unacceptable toxicity, or a maximum of 2 years. Treatment beyond progression is permitted in cases of oligoprogression amenable to local therapy.

Assessments Radiologic response assessments (CT ± CNS imaging) are performed every 6 weeks until week 12, then every 9 weeks until week 30, and every 12 weeks thereafter. HRQoL is assessed using NFLSI-17 and QLQ-ELD14 at baseline, every 6 weeks to week 12, every 9 weeks to week 30, and every 24 weeks thereafter.

Overall Treatment Utility (OTU) is assessed at the same intervals and incorporates:

* Radiological and clinical disease progression
* Toxicity profile and serious adverse events
* Patient-reported treatment acceptability Geriatric-specific assessments (hand-grip strength and timed up-and-go) are performed at baseline, week 12, week 30, and every 24 weeks.

Statistical Considerations With 128 OS events, the study is powered (80%) to detect an increase in median OS from 10.3 months (based on IPSOS trial) to 16 months in the experimental arm (one-sided alpha = 0.05). Sample size: 156 patients (allowing 5% attrition).

Time-to-event outcomes will be analyzed using Kaplan-Meier methods with log-rank tests and Cox proportional hazards models. Response rates and adverse events will be compared using Fisher's exact or chi-square tests. Continuous variables (e.g., HRQoL scores) will be analyzed using Wilcoxon rank-sum or linear regression (mixed models as appropriate).

Quality Assurance and Data Integrity

Although not formally a registry, the trial employs registry-like quality control elements:

* Data validation: Real-time data entry into electronic case report forms (eCRFs) with predefined logic and range checks.
* Source Data Verification (SDV): Conducted to ensure data accuracy and completeness via comparison with medical records and source documents.
* Standard Operating Procedures: SOPs are implemented, which cover all trial operations-site initiation, data collection, patient assessments, safety reporting, and amendment handling.
* Monitoring and auditing: Central and on-site monitoring according to a risk-based monitoring plan. Sites may be audited for compliance with ICH-GCP.
* Missing data management: Missing values due to dropout, nonresponse, or data inconsistency will be handled using pre-specified strategies, including sensitivity analyses.

Conclusion This trial responds to the pressing need for evidence-based, tolerable, and effective treatment strategies for older and/or frail patients with advanced NSCLC. By leveraging geriatric screening tools and integrating real-world adaptations such as reduced-dose chemotherapy, this study aims to optimize oncologic outcomes while preserving quality of life and functional status. Findings will inform clinical decision-making for a frequently excluded patient group in oncology research.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Histologically or cytologically confirmed NSCLC. Mixed histology with small-cell component is not allowed.
* Metastatic or advanced or recurrent NSCLC without a curative-intent treatment option (surgery or chemo-radiotherapy).
* PD-L1 <50% by local testing (SP 142 excluded)
* ≥70 years
* ECOG 0-2
* G8 screening score of ≤14 and/or ineligible for full-dose chemotherapy, defined as doses of carboplatin AUC 5, pemetrexed 500 mg/m2, paclitaxel 175 mg/m2, gemcitabine 1200 mg/m2 (as per Investigator)
* Life expectancy ≥6 months
* Patients with a prior malignancy (except NSCLC, see EC 7.2.2 and 7.2.3) and treated with curative intent are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of disease at registration. Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence, after consultation with CI.
* Patients with asymptomatic untreated or symptomatic treated CNS metastases are eligible if corticosteroid dose <10 mg prednisolone equivalent/day for at least 7 days
* Patients must be suitable to receive reduced-dose carboplatin-doublet chemotherapy in combination with immunotherapy including adequate bone marrow, renal and hepatic function as follows:

  * Hemoglobin ≥90 g/L, neutrophils ≥1.5 G/L, Thrombocytes ≥100G/L
  * Creatinine clearance (Cockroft-Gault) ≥30 mL/min
  * ASAT/ALAT ≤2xULN, Bilirubin ≤1.5xULN (≤3xULN for patients with Gilbert's disease),
* Men agree not to donate sperm or father a child during trial treatment and until 6 months after the last dose of trial treatment

Exclusion Criteria:

* Actionable genomic alteration for 1L treatment (EGFR, ALK, ROS1, RET, NTRK, MET Exon14 skipping). Testing is required for any NSQ-NSCLC or patients with SCC and a smoking history of ≤10py.
* Prior systemic treatment for metastatic NSCLC.
* Prior chemotherapy and/or immunotherapy in curative-intent treatment for locally advanced NSCLC in the past 6 months.
* Oligometastatic treatment concept with induction systemic therapy and planned LAT to all lesions.
* High tumor burden with a risk of rapid critical progression, as judged by the Investigator. Careful patient selection is important in order to prevent that patients in the comparator arm are not eligible for receiving add-on reduced-dose chemotherapy anymore if primary progression occurs (e.g., pericardial infiltration, high liver metastasis load etc).
* Active, treatment-requiring auto-immune disease in the past 2 years other than vitiligo, alopecia, hypothyroidism, type 1 diabetes or diet-controlled celiac disease.
* History of pneumonitis in the past 5 years.
* Systemic corticosteroid treatment ≥10 mg/day of prednisolone-equivalent or any other systemic immunosuppressive medication within 7 days prior to first dose of study intervention (except as needed for chemotherapy premedication or for physiologic corticosteroid replacement)
* Any infection requiring hospitalization or treatment with IV anti-infectives within 2 weeks of first dose of study medication
* Uncontrolled infection with HIV, hepatitis B or hepatitis C infection
* Receipt of a live vaccine within 4 weeks of start of study medication
* Receipt of COVID-19 vaccination within 1 week of planned start of study medication or for which the planned COVID-19 vaccinations would not be completed 1 week prior to start of study medication
* Organ transplant

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of randomization until the date of death from any cause, assessed up to 1 year after end of treatment.
  OS is defined as time from randomization to death due to any cause. Patients not experiencing an event will be censored at their last date known alive.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization until the date of confirmed tumor progression according to RECIST 1.1 or death from any cause, assessed up to 1 year after end of treatment.
  PFS is defined as time from randomization to confirmed tumor progression according to RECIST 1.1 or death due to any cause. Patients not experiencing an event will be censored at their last tumor assessment before starting a new anti-cancer treatment line (if any).
Objective response rate (ORR) | From the date of randomization until the end of treatment, estimated up to 1 year after randomization.
  Objective response is defined as any complete response (CR) or partial response (PR) according to RECIST 1.1 criteria achieved during treatment. Patients without any tumor assessment or with non-evaluable response during treatment will be considered as failures for this endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Mauti, MD, Study Chair — CH - Kantonsspital Winterthur
Locations (16):
- Switzerland (16):
  - HFR Fribourg, Fribourg, Villars-sur-Glâne
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Inselspital, Bern
  - Kantonsspital Baselland, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Spital Thurgau AG - Kantonsspital Frauenfeld, Frauenfeld
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital Olten - Solothurner Spitäler, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hôpital du Valais - Sion, Sion
  - EOC Istituto Oncologico della Svizzera Italiana (IOSI), Viganello
  - Kantonsspital Winterthur, Winterthur
  - KSW Kantonsspital Winterthur, Winterthur
  - Stadtspital Zürich Triemli, Zurich